CLINICAL TRIAL: NCT00980850
Title: Open Label, Randomized, Parallel-Group, Multi-Centre Study to Evaluate the Safety, Tolerability and Immunogenicity of Baxter H1N1 Vaccine and GlaxoSmithKline H1N1 Vaccine in Children 6 Months to 12 Years of Age
Brief Title: Swine Flu (Novel Influenza A H1N1) Vaccine Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Andrew Pollard, University of Oxford
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2009/08 H1N1
Record Dates: First submitted 2009-09-18; First posted 2009-09-21 (Estimated); Last update posted 2013-05-09 (Estimated); Status verified 2013-05

CONDITIONS: Influenza
Keywords: Flu vaccine; H1N1 swine flu virus; Immunogenicity; Reactogenicity
MeSH Terms: conditions — Influenza, Human | interventions — pandemrix

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Groups A1 and A2 (Experimental): Baxter vaccine
  Interventions: Biological: Baxter Novel Influenza A H1N1 Whole Virus Vaccine
- Groups B1 and B2 (Experimental): GSK vaccine
  Interventions: Biological: GlaxoSmithKline Novel Influenza A H1N1 Split Virion Vaccine

INTERVENTIONS:
Biological: Baxter Novel Influenza A H1N1 Whole Virus Vaccine — Two 0.5 ml doses of vaccine given within 3 weeks interval
  Other Names: Celvapan
  Arms: Groups A1 and A2
Biological: GlaxoSmithKline Novel Influenza A H1N1 Split Virion Vaccine — Two 0.25 ml doses of vaccine given within 3 weeks interval
  Other Names: Pandemrix
  Arms: Groups B1 and B2

SUMMARY:
In the first half of this year a novel Influenza A H1N1 virus has resulted in an influenza pandemic. The United Kingdom has seen a particularly high incidence of disease. The highest rates of disease are being seen in young children. In anticipation of an influenza pandemic two vaccine manufacturers, Baxter and GlaxoSmithKline, have gained marketing authorization approval from the European Medicines Agency (EMEA) for a pandemic strain vaccine under the "mockup" dossier route based on limited clinical trial data for a candidate H5N1 vaccine. This "mockup" dossier route for pandemic influenza vaccines allows the submission of a core pandemic dossier during the interpandemic period, which results in the approval of a mockup pandemic vaccine. This is followed by a fast track approval of the pandemic vaccine based on the submission of the pandemic variation when the situation arises. The Baxter and GlaxoSmithKline vaccines have now been modified to cover the novel influenza A H1N1 strain.

Given the high rates of swine flu disease in children, this age group is likely to particularly benefit from immunization against this virus, however there are few data on the use of these vaccines in a pediatric population. The proposed study therefore aims to assess the immunogenicity, safety, and tolerability of these two H1N1 vaccines when administered as two doses three weeks apart to children aged 6 months to 12 years of age.

DETAILED DESCRIPTION:
The study will be an open label, randomised, parallel group, multicentre clinical trial conducted by a consortium of the leading paediatric vaccine research units in the United Kingdom. The study will recruit healthy children 6 months to 12 years of age. Children with previously laboratory confirmed infection with swine flu will be excluded, as will those that have received a treatment course of oseltamivir. Children with immune deficiencies and egg allergy will also be excluded.

The study will be conducted as a collaboration between the Health Protection Agency and the following study recruitment sites: Oxford Vaccine Group (OVG), Bristol Children's Vaccine Centre (BCVC), the Royal Devon and Exeter Hospital, St George's Vaccine Institute (SGVI) and the University of Southampton Wellcome Trust Clinical Research Facility (USWTCRF). Families in the area of these research sites will be notified of the study by methods including print and electronic media, posters and direct mail out via the child health computer departments. The study visits themselves will be conducted in locations such as hospital outpatients, GP surgeries, or schools. General practitioners will be informed of the study and all immunisations administered during the study, as will the relevant child health computer department.

Participants will be randomised on 1:1 basis to receive 2 doses of either of the H1N1 influenza vaccines being studied. These vaccines will be given 2-3 weeks apart and the blood tests will be taken at baseline and around 3 weeks after completion of the 2 dose immunisation course. If at the start of the trial there is clinical data or a recommendation from JCVI that supports the use of a half dose of either vaccine in children under 3 years of age, this will be used for this age group and the ethics committee will be informed of this change.

Participants' families will be given diary cards to record local and systemic reactions to the vaccines administered, as well as recording daily temperatures for the 7 days after receipt of the vaccines. They will be telephoned 5-7 days after each vaccination to determine if there have been any SAEs since vaccination and to remind them to mail their completed diary cards to the HPA. Participants' families will also receive a memory card on which to record any visits to a doctor or emergency department from the 8th day after vaccine administration to the next study visit and any adverse events recorded in the diary card that are ongoing after day 7.

There will be 4 groups of children in the study:

Group A1: Children aged 6 months to less than 3 years of age will receive 2 doses of the Baxter H1N1 vaccine, 2-3 weeks apart. A blood sample will be taken at baseline and around 3 weeks after the second vaccine dose.

Group B1: Children aged 6 months to less than 3 years of age will receive 2 doses of the GSK H1N1 vaccine, 2-3 weeks apart. A blood sample will be taken at baseline and around 3 weeks after the second vaccine dose.

Group A2: Children aged greater than 3 years of age to 12 years of age will receive 2 doses of the Baxter H1N1 vaccine, 2-3 weeks apart. A blood sample will be taken at baseline and around 3 weeks after the second vaccine dose.

Group B2: Children aged greater than 3 years of age to 12 years of age will receive 2 doses of the GSK H1N1 vaccine, 2-3 weeks apart. A blood sample will be taken at baseline and around 3 weeks after the second vaccine dose.

ELIGIBILITY:
Inclusion Criteria:

* baby or child aged between 6 months to 12 years of age (i.e., to day before 13th birthday)
* for whom a parent/legal guardian has given written informed consent after the nature of the study has been explained
* available for all the visits scheduled in the study
* willingness to complete all study procedures

Exclusion Criteria:

* History of any vaccine against novel influenza A strain H1N1 (based on verbal confirmation from parent/guardian)
* Previous laboratory confirmed case of novel influenza A strain H1N1 or treatment with oseltamivir or zanamivir for novel influenza A strain H1N1 (n.b. a child commenced on treatment with oseltamivir or zanamivir for novel influenza A strain H1N1 whose treatment was stopped following negative microbiological tests for H1N1 on nasal swabs would be allowed to enrol in the study]
* History of severe allergic reaction after previous vaccinations or hypersensitivity to any H1N1 vaccine component
* Current egg allergy
* Known or suspected impairment/alteration of the immune system
* Disorders of coagulation
* Immunosuppressive therapy, use of systemic corticosteroids for more than 1 week within the 3 months prior to enrollment
* Receipt of blood, blood products and/or plasma derivatives or any immunoglobulin preparation within 3 months prior to enrollment
* Intent to immunize with any other vaccine(s) against novel influenza A strain H1N1 throughout the study period
* Participation in another clinical trial of an investigational medical product
* Any condition which, in the opinion of the investigator, might interfere with the evaluation of the study objectives. Children with chronic, stable medical illnesses that do not result in immunosuppression (e.g., cerebral palsy, epilepsy, cystic fibrosis, congenital heart disease) will be allowed to participate in the study, unless these conditions will in some way interfere with the completion of study procedures. Children with conditions that may alter the immune response to vaccines (e.g., Trisomy 21) or will affect the ability to accurately describe adverse events (e.g., children over 5 years of age but with severe learning difficulties) will be excluded

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1000 (Estimated)
Dates: Start 2009-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with a 4 fold rise in MN titre between the pre-vaccination sample and sample taken 3 weeks after the second dose | 3 weeks after second vaccine dose
Percentage of participants experiencing each of fever (≥ 38°C per axilla), local tenderness, local swelling or local erythema within the 7 days following each immunisation with the study vaccines | Within the 7 days following each immunisation with the study vaccines

SECONDARY OUTCOMES:
Percentage of subjects with an HAI titre ≥ 1 in 32 | 3 weeks after the second dose
Percentage of subjects with a 4 fold rise in HAI titre between the pre-vaccination sample and sample taken 3 weeks after the second dose | 3 weeks after the second dose
The geometric mean fold rises in HAI titres from baseline to after three weeks after 2 doses of the Baxter H1N1 vaccine and the GSK H1N1 vaccine. | 3 weeks after the second dose
The geometric mean fold rises in MN titres from baseline to three weeks after 2 doses of the Baxter H1N1 vaccine and the GSK H1N1 vaccine. | 3 weeks after the second dose
The geometric mean HAI and MN titres three weeks after 2 doses of the Baxter H1N1 vaccine and the GSK H1N1 vaccine. | 3 weeks after the second dose
Percentage of participants experiencing each of: reduced feeding, reduced activity, irritability, persistent crying, vomiting or diarrhoea, receiving medication for pain or temperature (6 month to 5 year olds). | Up to 3 weeks after the second dose
Percentage of participants experiencing each of: malaise, headache, nausea/ vomiting, diarrhoea, reduced appetite, muscle pain or joint pain, receiving analgesic/ antipyretic medication (5 to 12 year olds). | Up to 3 weeks after the second dose
The effect of genetic polymorphisms on the immunogenicity and reactogenicity of the H1N1 vaccines. | Up to 3 weeks after the second dose

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Pollard, MRCP, PhD, Study Director — Oxford Vaccine Group, University of Oxford; Liz Miller, FRCPath, DSc, Principal Investigator — Public Health England; Paul Heath, FRCPCH, Principal Investigator — St Georges Vaccine Institute; Adam Finn, PhD, FRCPCH, Principal Investigator — Bristol Children's Vaccine Centre; Saul Faust, MRCPCH, PhD, Principal Investigator — University of Southampton Wellcome Trust Clinical Research Facility; Andrew Collinson, MRCPCH, MD, Principal Investigator — Royal Devon and Exeter NHS Foundation Trust; Matthew Snape, FRCPCH, MD, Principal Investigator — Oxford Vaccine Group
Locations (5):
- United Kingdom (5):
  - Bristol Children's Vaccine Centre, Bristol, Bristol
  - St Georges Vaccine Institute, London, London
  - Royal Devon and Exeter NHS Foundation Trust, Exeter
  - Oxford Vaccine Group, Oxford
  - University of Southampton Wellcome Trust Clinical Research Facility, Southampton

REFERENCES:
- [Background] Andrews NJ, Walker WT, Finn A, Heath PT, Collinson AC, Pollard AJ, Snape MD, Faust SN, Waight PA, Hoschler K, Sheasby L, Waddington C, Kerridge S, Chalk J, Reiner A, John T, Fletcher M, Allen R, Fineman N, Wilkins S, Casey M, Michaelis L, Oeser C, Okike I, Ladhani S, Miller E. Predictors of immune response and reactogenicity to AS03B-adjuvanted split virion and non-adjuvanted whole virion H1N1 (2009) pandemic influenza vaccines. Vaccine. 2011 Oct 19;29(45):7913-9. doi: 10.1016/j.vaccine.2011.08.076. Epub 2011 Aug 27. PMID 21875635
- [Background] Waddington CS, Walker WT, Oeser C, Reiner A, John T, Wilkins S, Casey M, Eccleston PE, Allen RJ, Okike I, Ladhani S, Sheasby E, Hoschler K, Andrews N, Waight P, Collinson AC, Heath PT, Finn A, Faust SN, Snape MD, Miller E, Pollard AJ. Safety and immunogenicity of AS03B adjuvanted split virion versus non-adjuvanted whole virion H1N1 influenza vaccine in UK children aged 6 months-12 years: open label, randomised, parallel group, multicentre study. BMJ. 2010 May 27;340:c2649. doi: 10.1136/bmj.c2649. PMID 20508026
- [Background] Waddington C, Andrews N, Hoschler K, Walker W, Oeser C, Reiner A, John T, Wilkins S, Casey M, Eccleston P, Allen R, Okike I, Ladhani S, Sheasby E, Waight P, Collinson A, Heath P, Finn A, Faust S, Snape M, Miller E, Pollard A. Open-label, randomised, parallel-group, multicentre study to evaluate the safety, tolerability and immunogenicity of an AS03(B)/oil-in-water emulsion-adjuvanted (AS03(B)) split-virion versus non-adjuvanted whole-virion H1N1 influenza vaccine in UK children 6 months to 12 years of age. Health Technol Assess. 2010 Oct;14(46):1-130. doi: 10.3310/hta14460-01. PMID 20923610